CLINICAL TRIAL: NCT05886582
Title: Phase 2a Double-Blind Placebo-Controlled Trial of Transdermal Rotigotine as Adjunct to Behavioral Therapy for Cocaine Use Disorder
Brief Title: Transdermal Rotigotine as Adjunct to Behavioral Therapy for Cocaine Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20026910; 1U01DA057846-01 (NIH)
Record Dates: First submitted 2023-04-27; First posted 2023-06-02 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Rotigotine (RTG) (Experimental): Participants who are randomized to the active RTG arm will receive Neupro® RTG patches
  Interventions: Drug: Rotigotine Transdermal System [Neupro]
- Placebo (Placebo Comparator): Participants who are randomized to placebo will receive transdermal patches that match the size and color of active Neupro®.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine Transdermal System [Neupro] — Neupro® 2mg/24h transdermal patches for the first seven days, followed by the target 4mg dose for the subsequent 35 days (five weeks) of dosing up to the follow-up assessments, followed by two days of 2mg/24h ramp-down dose.
  Arms: Active Rotigotine (RTG)
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 2b pilot clinical trial to determine whether non-ergoline D3/D2/D1 dopamine (DA) receptor agonist rotigotine (RTG), in combination with treatment as usual, including individual or group behavioral therapy can a) reduce cocaine use and also b) increase brain activity in frontocortical areas of the brain, and, as a reflection of that - improve top-down cognitive control in persons with cocaine use disorder (CocUD).

Rotigotine is a marketed non-ergoline D3/D2/D1 DA agonist (RTG, Neupro®) in the form of a transdermal patch that is FDA-approved for the treatment of Parkinson's Disease and Restless Legs Syndrome. The premise of this project was based on apparent beneficial effects of RTG in a different human population characterized by executive function (EF) impairment. In light of the deficits in EF common in persons with CocUD, RTG may hold the potential for cognitive improvement in persons with CocUD who are in treatment as usual to both attend to and retain psychoeducation concepts better. In addition, rotigotine may help these individuals in recovery maintain goals better, where goal maintenance is a crucial integrative product of successful EF.

DETAILED DESCRIPTION:
Among different substance use disorders, stimulant use disorders are more consistently linked with impaired executive function (EF) of the brain, which is a set of cognitive skills like working memory that operate to enable self-control over behavior and long-term planning. Medications such as stimulants that increase function of the frontal cortex dopamine (DA) system can improve EF. However, stimulants such as amphetamine have abuse potential. Of interest is determining whether a multiple DA receptor medication like rotigotine could improve brain function in persons with stimulant use disorder who are in therapy, to help them retain educational concepts and strategies better. Rotigotine has been shown to improve cognition-related quality of life in persons with Alzheimer's Disease. This is a roughly six week trial of rotigotine (given in a skin patch) to determine whether it not only reduces cocaine use in persons in treatment for cocaine use disorder, but actually improves cognitive performance itself, and increases activity in the frontal cortex of the brain, compared to placebo. It is hypothesized that rotigotine will be specifically helpful for cognition and abstinence in those participants whose cognitive performance ability tested at baseline is below the median.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 25 and 70 years of age.
* Meet current DSM-5 criteria for Cocaine Use Disorder (CocUD), moderate or severe
* Able to understand and comply with study procedures
* Have positive urine result for cocaine metabolite benzoylecgonine (BE) during at least one screening visit (out of up to three visits, depending on participants' preference) AND/OR self-report of recent cocaine use (approximately past 30 days).
* Have hematology and chemistry laboratory tests that are within normal limits, except that liver function tests must be no more than 2x of the upper limit of normal (if any elevation is above the limit - must be judged by the study physician to be clinically insignificant).
* No clinically significant abnormalities on baseline ECG.
* Be able to demonstrate an understanding of study procedures and follow instructions including behavioral laboratory and fMRI testing.
* Women must either be unable to conceive (i.e., surgically sterilized, sterile, or postmenopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device with spermicide, or condoms). Men will be advised to use condoms. All females must provide negative pregnancy urine tests before study entry, at each visit during the study, and the end of study participation.
* Body Mass Index (BMI) between 18-45kg/M2 and weight of at least 50kg at screening

Exclusion Criteria:

* Have concurrent secondary DSM-5 diagnosis of any psychoactive substance use disorder other than cocaine, alcohol, methamphetamine, nicotine, opioid, or marijuana use disorder.
* Have a DSM-5 axis I psychiatric disorder other than substance use disorder, including but not limited to Bipolar I Disorder, Schizophrenia, or other psychotic disorder that require treatment with antipsychotics, or a neurological disorder requiring ongoing treatment and/or making study participation unsafe. Comorbid PTSD, Generalized Anxiety Disorder and Major Depressive Disorder will be allowed.
* Consistent and regular (as opposed to intermittent, infrequent, or as needed) use of medications contraindicated for concurrent use along with RTG, or would confound the mechanism of RTG action and data interpretation. These include DA antagonists such as antipsychotic medications (especially neuroleptics) or metoclopramide.
* Subjects with evidence or history of any clinically significant medical disorder including biliary obstruction, clinically significant hepatic disease, severe cardiovascular or pulmonary disease, bronchial asthma, renal, or endocrine disease. However, controlled hypertension, controlled hypothyroidism, and cancer in remission over 5 years will not be excluded.
* Have a history of seizures (excluding childhood febrile seizures) or loss of consciousness (e.g. from traumatic brain injury) for more than 30 minutes.
* Have significant current suicidal or homicidal ideation or a suicide attempt within the past 6 months, based on the Columbia Suicide Severity Rating Scale (C-SSRS).
* Be HIV positive by self-report or history.
* Be pregnant or nursing or not using a reliable form of contraception if able to conceive. All females must provide negative pregnancy urine tests before study entry, at each visit during the study, and the end of study participation
* Have any other illness, or condition, which in the opinion of the clinical co-investigator (Arias) would preclude safe and/or successful completion of the study.
* Be allergic to rotigotine.
* Have taken any investigational drug within 45 days prior to baseline
* Demonstrate intolerance to, poor adherence to, or extreme skin irritation by daily application of known placebo "practice" skin patches during the screening phase
* Current/pending criminal charges that may result in incarceration within the next 60 days
* Self-report of allergic or other reactions to sulfites (e.g. in foods)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cocaine-positive urine samples | weeks 5 - 6 of transdermal patch treatment
  comparison of cocaine-positive urine samples between participants randomized to transdermal RTG relative to participants randomized to placebo patches
self-reported cocaine use | weeks 5 - 6 of transdermal patch treatment
  comparison of cocaine cocaine use (by self report) between participants randomized to transdermal RTG relative to participants randomized to placebo patches

SECONDARY OUTCOMES:
executive function (change) | change from baseline to study week 6
  Change in CNS-VS Neurocognition Index (NCI) scores
QoLI total score (change) | change from baseline to study week 6
  Change in QoLI total scores
dorsolateral prefrontal cortex (DLPFC) | study day 1 to study week 6
  Change in recruitment of dorsolateral prefrontal cortex (DLPFC)
stop signal task (SST) | study day 1 to study week 6
  Change in recruitment of right anterior insula by stop-signals in the SST
EC from DLPFC to striatum during working memory demands | study day 1 to study week 6
  change in EC from DLPFC to striatum during working memory demands in the EFNBk and during resting state

CONTACTS AND LOCATIONS:
Overall Officials: James M Bjork, PhD, Principal Investigator — Virginia Commonwealth University; Albert Arias, MD, Principal Investigator — Virginia Commonwealth University; Tanya Ramey, PHD, Study Director — National Institute on Drug Abuse (NIDA)
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No